CLINICAL TRIAL: NCT00840554
Title: The Effects of Adding a Home Exercise Program (HEP) to a Clinical Physical Therapy Program (CPTP) on the Cancer-Related Fatigue Reported by Patients Undergoing Concurrent Radiation and Chemotherapy for High-Grade Glioma (HGG)
Brief Title: The Effects of Adding a Home Exercise Program to a Clinical Physical Therapy Program on Cancer-Related Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HEP-001
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Fatigue
Keywords: Fatigue; Cancer-related fatigue; High grade glioma; Quality of life; Exercise; Physical Therapy; HGG; QOL
MeSH Terms: conditions — Fatigue; Glioma; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Therapy (Active Comparator)
  Interventions: Other: Clinic-based physical therapy program.
- Home Exercise (Experimental)
  Interventions: Other: Home exercise program.

INTERVENTIONS:
Other: Clinic-based physical therapy program. — All patients will receive a routine clinic-based physical therapy program. This program may include supervised aerobic conditioning, strengthening exercise, balance retraining, functional activity training, therapeutic exercise, and manual therapy.
  Other Names: PT
  Arms: Physical Therapy
Other: Home exercise program. — In addition to the clinic-based physical therapy program, patients will perform home exercises. Home exercise will include a walking and strengthening program 5 days per week. The home exercise routine will be recorded in an exercise diary.
  Other Names: Exercise
  Arms: Home Exercise

SUMMARY:
The purpose of this study is to find out if adding a home exercise program to a clinic physical therapy program will improve the fatigue experienced by patients being treated with concurrent chemotherapy and radiation therapy for high grade gliomas.

DETAILED DESCRIPTION:
Cancer-related fatigue is a common and disabling symptom in patients undergoing outpatient therapies to treat their cancers. Despite a consistent increase in both awareness and research, cancer-related fatigue remains poorly understood and poorly treated by the worldwide medical community.

The physical and emotional impact of cancer-related fatigue on Activities of Daily Living and Independent Activities of Daily Living can be profound. Simple tasks such as preparing meals and performing household chores become laborious. Walking up and down the aisles of grocery stores may send a patient directly to bed for the rest of the day upon returning home. In addition, if cancer-related fatigue contributes to prolonged bed rest, the secondary development of other medical problems can further impact quality of life and possibly length of life. Furthermore, the economic impact of cancer-related fatigue includes patients taking more days off work and reducing the number of hours they are able to work. Lastly, cancer-related fatigue often impacts the psychosocial well-being and family dynamics of patients, caregivers and their families.

Exercise is the strongest non-pharmacological intervention for management of cancer-related fatigue. Certain exercises have specifically demonstrated reduction in fatigue. An exercise program that incorporates strengthening and aerobic conditioning can decrease fatigue scores. Improvements in patient-reported cancer-related fatigue through the use of exercise has been demonstrated in various diseases, such as anemia, and several cancer types, most notably breast cancer. Furthermore, home exercise programs have shown meaningful improvements in patient reported fatigue.

This study will determine the effect that the addition of a 6-week Physical Therapist-directed home exercise program has on the pattern, severity, and quality of life of patient reported fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than 18 years old on day of enrollment, male or female.
2. Histological confirmation of a high grade glioma (HGG). The patient's treatment plan must include plans for concurrent radiation and chemotherapy at the University of Florida.
3. Patients otherwise meeting standard medical criteria for referral to physical therapy.
4. Physically capable of trial participation, defined as:

   * Ambulatory, without assist-devices.
   * Able to maintain a specified walking pace for 15-30 minutes.
5. Adequate medical health to participate in this study.
6. Absence of factors that have been documented to possibly confound the assessment of fatigue:

   * Hematocrit (Hct) <30.
   * Thyroid Stimulating Hormone (TSH) > 2.5 wnl.
7. Absence of other factors, such as inadequate nutritional level, pain control, electrolyte levels, depression, that are felt insufficient for trial participation.
8. Karnofsky Performance Status >60 or ECOG Performance Status <2.
9. Ability to read and understand the patient informed consent form.
10. Ability and willingness to follow all requirements of the study including following all directions, taking medication as prescribed, and completion of all diaries and forms.
11. Signed informed consent.

Exclusion Criteria:

1. Failure to meet inclusion criteria
2. Physical and medical issues that would interfere with trial participation, such as:

   * History of major cardiopulmonary symptoms.
   * Orthopedic problem limiting participation.
   * Dementia or poor mental status.
   * Neurological deficit limiting participation physically or cognitively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Determine the effect of a 6-week Physical Therapist-directed home exercise program on the pattern of patient reported fatigue. | 6 Weeks

SECONDARY OUTCOMES:
Determine the effect of a 6-week Physical Therapist-directed home exercise program on the severity of patient reported fatigue. | 6 Weeks
Determine the effect of a 6-week Physical Therapist-directed home exercise program on routine quality of life measurements and outcome. | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Erin M Dunbar, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States